CLINICAL TRIAL: NCT01285037
Title: A Phase 1 Study of LY2801653 in Patients With Advanced Cancer
Brief Title: A Study of LY2801653 in Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13008; I3O-MC-JSBA (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — merestinib; Cetuximab; Cisplatin; Gemcitabine; Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2801653 (Experimental): This study consists of a dose escalation of LY2801653 (Part A) followed by dose confirmation cohorts in four tumor types (adenocarcinoma of the colon or rectum, head and neck squamous cell carcinoma, uveal melanoma with liver metastasis, and cholangiocarcinoma) (Part B).
  Part C consists of dose determination for LY2801653 in combination with cetuximab in participants with head and neck squamous cell carcinoma followed by an expansion cohort.
  Part D consists of dose determination for LY2801653 in combination with cisplatin in participants with cholangiocarcinoma followed by an expansion cohort.
  Part E consists of dose determination for LY2801653 in combination with gemcitabine and cisplatin.
  Part F consists of dose determination for LY2801653 in combination with ramicirumab.
  Interventions: Drug: LY2801653; Drug: Cetuximab; Drug: Cisplatin; Drug: Gemcitabine; Drug: Ramucirumab

INTERVENTIONS:
Drug: LY2801653 — LY2801653 given orally once daily during 28-day cycles. Participants may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criterion is met.
Drug: Cetuximab — Cetuximab given via IV infusion once weekly, 400mg/m2 for first dose and 250mg /m2 for subsequent doses. If LY2801653 treatment is stopped due to toxicity after a minimum of 4 cycles, cetuximab may be continued until disease progression. In the event cetuximab treatment is stopped, participants may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criterion is met.
Drug: Cisplatin — Cisplatin given via IV infusion once a week for 2 weeks and then every 3 weeks. If the LY2801653 is terminated for LY2801653-related toxicity after a minimum of 4 cycles, cisplatin may be continued as monotherapy until progression of disease. Participants discontinuing cisplatin therapy may be allowed to continue single agent LY2801653 if they are receiving clinical benefit.
Drug: Gemcitabine — Gemcitabine given via IV infusion once a week for 2 weeks and then every 3 weeks. If the LY2801653 is terminated for LY2801653-related toxicity after a minimum of 4 cycles, gemcitabine may be continued as monotherapy until progression of disease. Participants discontinuing gemcitabine therapy may be allowed to continue single agent LY2801653 if they are receiving clinical benefit.
  Other Names: LY188011; Gemzar
Drug: Ramucirumab — Ramucirumab given via IV infusion every 2 weeks in a 28-day treatment cycle. Treatment with ramucirumab may continue until excessive toxicity or evidence of disease progression. In the absence of disease progression, treatment with LY2801653 may continue even if ramucirumab is discontinued provided no dose limiting toxicity related to LY2801653 is present. In the event that LY2801653 is discontinued, treatment with ramucirumab may be continued if there is no dose limiting toxicity related to ramucirumab.
  Other Names: IMC-1121B; LY3009806; Cyramza

SUMMARY:
Part A- The purpose of this study is to determine a safe dose of LY2801653 to be given to participants with advanced cancer and to determine any side effects that may be associated with LY2801653 in this participant population. Efficacy measures will be used to assess the activity of LY2801653.

Part B- The dose determined in Part A will be used along with efficacy measures to assess the activity of LY2801653 in participants with adenocarcinoma of the colon or rectum, head and neck squamous cell carcinoma (HNSCC), uveal melanoma with liver metastasis, and cholangiocarcinoma.

Part C - the objective of Part C is to determine a recommended Phase 2 dose of LY2801653 that may be safely given to participants with HNSCC when taken with standard doses of cetuximab Part D - the objective of Part D is to determine a recommended Phase 2 dose of LY2801653 that may be safely given to participants with cholangiocarcinoma when taken with a standard dose of cisplatin.

Part E - the objective of Part E is to determine a recommended Phase 2 dose of LY2801653 that may be safely given to participants with cholangiocarcinoma when taken with gemcitabine plus cisplatin.

Part F - the objective of Part F is to determine a recommended Phase 2 dose of LY2801653 that may be safely given to participants with gastric cancer when taken with ramucirumab.

DETAILED DESCRIPTION:
Parts C and D were added to the registration in November, 2013, per protocol amendment. Parts E and F were added to the registration in February, 2015, per protocol amendment.

ELIGIBILITY:
Inclusion Criteria:

* Part A- Diagnosed with advanced and/or metastatic cancer during dose escalation
* Part B- Diagnosed with adenocarcinoma of the colon or rectum, head and neck squamous cell carcinoma, uveal melanoma with liver with metastasis, or cholangiocarcinoma
* Part C - Diagnosed with head and neck squamous cell carcinoma and have received at least one prior platinum-based systemic therapy
* Part D - Diagnosed with cholangiocarcinoma and have not received more than 1 prior systemic therapy
* Part E - Diagnosed with cholangiocarcinoma, either intrahepatic or extrahepatic, that is unresectable, recurrent, or metastatic. Participants must not have received prior systemic front line therapy for metastatic or resectable disease (i.e. participants may have received adjuvant gemcitabine but have not yet received gemcitabine/cisplatin for recurrent metastatic disease). Participants must be, in the opinion of the investigator, an appropriate candidate for experimental therapy. Participants should be evaluated for the need to undergo biliary drainage by stent placement prior to study participation. Participants should have adequate biliary drainage with no unresolved biliary obstruction.
* Part F - Histologically- or cytologically-confirmed gastric carcinoma, including gastric adenocarcinoma or gastroesophageal junction (GEJ) adenocarcinoma (participants with adenocarcinoma of the distal esophagus are eligible if the primary tumor involves the GEJ). Participants must be ramucirumab naïve. Participants must be, in the opinion of the investigator, an appropriate candidate for experimental therapy. human epidermal growth factor receptor 2 (HER2)/neu status should be documented, if known.
* Must be at least 18 years of age
* Adequate hematologic, renal, and liver functions
* Eastern Cooperative Oncology Group (ECOG) status of 0 or 1
* Ability to swallow capsules, with the exception of head and neck squamous cell carcinoma participants who may have study drug crushed and administered through a feeding tube

Exclusion Criteria:

* Have serious preexisting medical conditions that would preclude participation in the study
* Have a chronic underlying infection
* Have symptomatic central nervous system (CNS) malignancy or metastasis
* Have current acute or chronic leukemia
* Are pregnant or lactating
* Have hepatocellular cancer, liver cirrhosis with a Child-Pugh stage of B or higher, or have received a liver transplant
* Have a history of congestive heart failure with a New York Heart Association class greater than 2, unstable angina, recent myocardial infarction (within 6 months of study enrollment), transient ischemic attacks, stroke, or arterial or venous vascular disease
* Have a QTc interval greater than 470 msec
* For participants in Part B, C, D, E, and F, a tumor tissue sample is mandatory, when safe and feasible, for biomarker analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2009-09-09 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2017-09-11 (Actual)

PRIMARY OUTCOMES:
Recommended dose for phase 2 studies: Maximum tolerated dose | Baseline to study completion (estimated as 3 months)

SECONDARY OUTCOMES:
Number of participants with tumor response | Part A: Baseline to study completion (estimated as 3 months)
Clinical benefit rate (CBR) | Parts B, C, D: Baseline to study completion (estimated as 3 months)
Progression free survival (PFS) | Parts B, C, D: Baseline to study completion (estimated as up to 6 months)
Duration of response | Parts B, C, D: Baseline to study completion (estimated as up to 6 months)
Number of participants with clinically significant effects | Baseline to study completion (estimated as 3 months)
Pharmacokinetics: Area under the concentration/time curve (AUC) | Cycle 1, Day 1; Cycle 2, Day 1
Pharmacokinetics: Maximum plasma concentration (Cmax) | Cycle 1, Day 1; Cycle 2, Day 1
Maximum tolerated dose (MTD) of LY2801653 in combination with cetuximab for phase 2 studies in HNSCC | Baseline to study completion (estimated as 3 months)
Maximum tolerated dose (MTD) of LY2801653 in combination with cisplatin for phase 2 studies in cholangiocarcinoma | Baseline to study completion (estimated as 3 months)
Maximum tolerated dose (MTD) of LY2801653 in combination with gemcitabine plus cisplatin for phase 2 studies in cholangiocarcinoma | Baseline to study completion (estimated as 3 months)
Maximum tolerated dose (MTD) of LY2801653 in combination with ramucirumab for phase 2 studies in gastric carcinoma | Baseline to study completion (estimated as 3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-817-285-4559) or 1-317-615-4559 Mon - Fri 9AM to 5PM Eastern time (UTC/GMT - 5hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- United States (7):
  - Arizona Cancer Center, Tucson, Arizona
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Mount Sinai Medical Center, New York, New York
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] He AR, Cohen RB, Denlinger CS, Sama A, Birnbaum A, Hwang J, Sato T, Lewis N, Mynderse M, Niland M, Giles J, Wallin J, Moser B, Zhang W, Walgren R, Plimack ER. First-in-Human Phase I Study of Merestinib, an Oral Multikinase Inhibitor, in Patients with Advanced Cancer. Oncologist. 2019 Sep;24(9):e930-e942. doi: 10.1634/theoncologist.2018-0411. Epub 2019 Mar 4. PMID 30833489
- [Derived] Yan SB, Peek VL, Ajamie R, Buchanan SG, Graff JR, Heidler SA, Hui YH, Huss KL, Konicek BW, Manro JR, Shih C, Stewart JA, Stewart TR, Stout SL, Uhlik MT, Um SL, Wang Y, Wu W, Yan L, Yang WJ, Zhong B, Walgren RA. LY2801653 is an orally bioavailable multi-kinase inhibitor with potent activity against MET, MST1R, and other oncoproteins, and displays anti-tumor activities in mouse xenograft models. Invest New Drugs. 2013 Aug;31(4):833-44. doi: 10.1007/s10637-012-9912-9. Epub 2012 Dec 29. PMID 23275061
- See also: Click here for more information about this study:A Study of LY2801653 in Participants With Advanced Cancer — https://www.lillytrialguide.com/en-US/studies/stomach-cancer/JSBA#?postal=